CLINICAL TRIAL: NCT02640989
Title: Safety and Immunogenicity of Three Seasonal Trivalent Influenza Vaccines in China Military
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Center for Disease Prevention and Control of Beijing Military Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-INF-BJJQ-01
Record Dates: First submitted 2015-12-04; First posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Influenza
Keywords: Influenza Vaccine; Safety; Immunogenicity
MeSH Terms: conditions — Influenza, Human | interventions — vaxigrip; fluarix

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): * Single intramuscular injection of the investigational vaccine (0.5 ml) on Day 0
  * Seasonal trivalent influenza vaccine, Anflu®
  Interventions: Biological: Seasonal trivalent influenza vaccine, Anflu®
- Group 2 (Experimental): * Single intramuscular injection of the investigational vaccine (0.5 ml) on Day 0
  * Seasonal trivalent influenza vaccine, VAXIGRIP
  Interventions: Biological: Seasonal trivalent influenza vaccine, VAXIGRIP
- Group 3 (Active Comparator): * Single intramuscular injection of the investigational vaccine (0.5 ml) on Day 0
  * Seasonal trivalent influenza vaccine, Fluarix
  Interventions: Biological: Seasonal trivalent influenza vaccine, Fluarix

INTERVENTIONS:
Biological: Seasonal trivalent influenza vaccine, Anflu® — Seasonal trivalent influenza vaccine manufactured by Sinovac Co., Ltd.
  Other Names: Anflu®
  Arms: Group 1
Biological: Seasonal trivalent influenza vaccine, VAXIGRIP — Seasonal trivalent influenza vaccine manufactured by PasteurSanofi Pasteur
  Other Names: VAXIGRIP
  Arms: Group 2
Biological: Seasonal trivalent influenza vaccine, Fluarix — Seasonal trivalent influenza vaccine manufactured by GlaxoSmithKline Biologicals
  Other Names: Fluarix
  Arms: Group 3

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of three seasonal trivalent influenza vaccines (TIVs)manufactured by Glaxosmith Kline (GSK), Beijing Sinovac Biotech (Sinovac) and Shenzhen Sanofi Pasteur (Pasteur) in Chinese healthy servicemen. Using imported GSK's TIV as control, to compare it with other two domestic TIVs in Chinese healthy servicemen.

DETAILED DESCRIPTION:
This study is a 1:1:1 randomized, double-blinded, controlled phase Ⅳ clinical trial in a military command in Beijing. Healthy individuals aged between 18～34 years who had not received any influenza vaccine during recent three years will be enrolled and administrated one dose TIV. Safety data will be collected for whole study (Day 0 to Day 30).Blood samples will be collected for immunogenicity assessments before injection and 21 days after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy servicemen aged between 18-34 years ,who had not received any influenza vaccine during recent three years;
* Proven legal identity;
* Written informed consent;
* Complying with the requirement of the study protocol;

Exclusion Criteria:

* Pregnant, breast feeding women;
* History of allergy to any vaccine or vaccine ingredient;
* Receipt of any immunosuppressant within 6 month prior to study entry;
* Congenital malformation, developmental disorders, serious chronic diseases, autoimmune disease, immunodeficiency, serious cardiovascular disease, diabetes, Guillain-Barré syndrome, hypertension that cannot be stabilized by medication, liver or kidney disease, or malignant tumor;
* Acute disease or acute stage of chronic disease within 7 days prior to study entry;
* Axillaty temperature > 37.0 °C;
* Any other factor that in the opinion of the investigator suggesting the volunteer is unsuitable for this study;

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 292 (Actual)
Dates: Start 2014-10; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Hemagglutination inhibition (HI) titers of each strain which were recommended by WHO for the 2014 seasonal influenza vaccines | 21 days after vaccination
  Hemagglutination inhibition (HI) titers were measured using the antigen and standard serum provided by the National Institute for Biological Standards and Control (NIBSC).

SECONDARY OUTCOMES:
The incidences of adverse events (AEs) | 21 days after vaccination
  After vaccination, occurrences of AEs were collected till day 21. Each AE case was reviewed by the investigator to determine whether or not it was an adverse reaction (related to the vaccination).
The post-vaccination seroprotection rates of each of the influenza vaccines | 21 days after vaccination
  Hemagglutination inhibition (HI) titers were used to calculate post-vaccination seroprotection rates of each of the influenza vaccines. By European Committee(European criteria): in adults aged between 18 to 60, post-vaccination seroprotection rates should be ≥ 70% for all vaccine strains.
The post-vaccination seroconversion rates of each of the influenza vaccines | 21 days after vaccination
  Hemagglutination inhibition (HI) titers were used to calculate post-vaccination seroconversion rates of each of the influenza vaccines. By European Committee(European criteria): in adults aged between 18 to 60, post-vaccination seroconversion rates should be > 40% for all vaccine strains.
The post-vaccination mean geometric increases (GMIs) of each of the influenza vaccines | 21 days after vaccination
  Hemagglutination inhibition (HI) titers were used to calculate post-vaccination mean geometric increases (GMIs) of each of the influenza vaccines. By European Committee(European criteria): in adults aged between 18 to 60, post-vaccination mean geometric increases (GMIs) should be ≥ 2.5 for all vaccine strains.

CONTACTS AND LOCATIONS:
Overall Officials: Dongqi Gao, PhD, Principal Investigator — Center for Disease Prevention and Control of Beijing Military Region
Locations (1):
- Center for Disease Prevention and Control of Beijing Military Region, Beijing, Beijing Municipality, China